CLINICAL TRIAL: NCT06578754
Title: Validation Test for Plasma Oxalate Level in a Biochemical Laboratory at the Galilee Medical Center
Brief Title: Validation Testing for Plasma Oxalate Levels in the Biochemical Laboratory at the Galilee Medical Center, in Collaboration With the Biochemistry Laboratory at CHARITE Hospital in Berlin, and Testing the Relationship Between Oxalate Levels and Vitamin C Levels in Plasma
Status: Not yet recruiting | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Hadas Shasha-Lavsky, Principle Investigator, Western Galilee Hospital-Nahariya
Other Study IDs: 0096-24-NHR
Record Dates: First submitted 2024-08-20; First posted 2024-08-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hyperoxaluria
Keywords: plasma oxalate level, hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy volunteers: About 10 blood samples to be taken from this group
  Interventions: Other: This is an non-interventional study
- Dialysis patients without a background of hyperoxaluria: About 10 blood samples to be taken from this group as well as 20 additional blood samples from dialysis patients where oxalate levels and vitamin C levels will be tested
  Interventions: Other: This is an non-interventional study
- Hyperoxaluria patients receiving drug treatment or after a liver transplant: About 5 blood samples from this group
  Interventions: Other: This is an non-interventional study
- Patients advanced kidney failure not on dialysis: About 5 blood samples from this group
  Interventions: Other: This is an non-interventional study

INTERVENTIONS:
Other: This is an non-interventional study — Only blood samples will be required in this study. It is noninterventional.

SUMMARY:
Background:

Elevated plasma oxalate levels in various conditions, including: primary hyperoxaluria due to increased production in the liver, renal failure due to decreased renal excretion, intestinal diseases with fatty diarrhea due to increased intestinal absorption, and increased intake of substances containing oxalate or sources of oxalate. Primary hyperoxaluria type 1 is a rare hereditary disease in which there is an increase in oxalate production in the liver due to a defect in the AGT enzyme in the oxalate metabolism pathway. The disease causes end-stage renal failure, and until recently, the only treatment was liver and kidney transplantation. The disease is more common in our region, and the Pediatric Nephrology Unit is a center of expertise for this disease. In 2022, a new treatment for hyperoxaluria type 1, which is an alternative to liver transplantation (Lomecirane), was added to the health basket. With the introduction of this treatment in Israel, there was a need to test the level of oxalate in plasma in order to monitor the response to treatment and as part of the preparation for kidney transplantation in cases of type 1 hyperoxaluria with end-stage renal failure. There is no laboratory in Israel that performs plasma oxalate testing. The biochemistry laboratory at the Galilee Medical Center performs oxalate testing in urine using an enzymatic method. Testing for oxalate in plasma using this method requires external validation because the manufacturer intends this test for urine only. There are laboratories around the world that use this method to measure oxalate in plasma.

Vitamin C is a precursor (source) for oxalate in the body. High vitamin C levels in dialysis may lead to increased oxalate, which is associated with worsening kidney damage and damage to other organs, including an increase in the incidence of cardiovascular disease. Dialysis patients are therefore advised to avoid vitamin C supplements. On the other hand, cases of symptomatic vitamin C deficiency in dialysis patients have been described due to their tendency to have an inadequate diet. One case was described in the literature by the Nephrology Department at our institution.

Objectives:

1. To validate the plasma oxalate test by comparing it to an external laboratory that performs the test.
2. To examine the relationship between vitamin C levels and plasma oxalate levels in patients with varying degrees of renal failure.

Importance:

1. Establishment of a laboratory service that does not currently exist in Israel and is clinically important for treatment decisions.
2. Assessing the relationship between vitamin C levels and oxalate levels in renal failure will help in the tailored treatment of these patients and prevent complications of vitamin C deficiency on the one hand or hyperoxaluria secondary to vitamin C excess on the other.

DETAILED DESCRIPTION:
Background:

The source of oxalate in the body is endogenous production in the liver and diet. Oxalate is excreted in the urine by the kidneys. In situations where there is excess oxalate in the urine, it may crystallize together with calcium and settle as calcium oxalate crystals in the kidney, causing kidney damage. In cases of advanced kidney damage, oxalate excretion in urine is impaired, and oxalate accumulates in the blood and precipitates in all tissues of the body, including the eyes, bones, bone marrow, blood vessels, and more. Conditions in which there are high levels of oxalate in the body are caused by poisoning (e.g., ethylene glycol) or secondary hyperoxaluria conditions such as cystic fibrosis or inflammatory bowel disease (there is increased oxalate absorption in the intestine in cases of fatty diarrhea) or primary hyperoxaluria.

Hyperoxaluria is a group of diseases caused by increased oxalate secretion by the liver due to a genetic defect in the oxalate metabolism pathway in the liver. Type 1 hyperoxaluria (PH1) is the most severe of the group, causing kidney failure in most patients by the second decade of life. Until recently, treatment for PH1 was based on liver transplantation to restore normal enzyme function, and in most cases, kidney transplantation was also required1. In November 2021, the FDA approved a breakthrough drug for hyperoxaluria, LUMASIRAN2.

There are a number of laboratories, including the biochemistry laboratory at the Galilee Medical Center, that perform urine oxalate level testing. The urine test is performed as an initial screening in situations where hyperoxaluria is suspected, as part of the investigation of kidney stones, and as a follow-up to the response to the new PH1 drug treatment.

The Pediatric Nephrology Unit at the Galilee Medical Center is a center of expertise for hyperoxaluria. The incidence of this disease in the Galilee population is among the highest in the world, and as a result, our center has accumulated extensive experience in treating this disease.

In addition, the Pediatric Nephrology Unit served as a center for ALNYLAM's clinical research to test the efficacy and safety of the drug LUMASIRAN. Currently, there are eight PH1 patients receiving the new drug who are being monitored by the Pediatric Nephrology Unit at our institution.

Plasma oxalate testing is mainly required in cases of primary hyperoxaluria, to monitor response to treatment, in preparation for kidney transplantation, and as follow-up after kidney transplantation. There are other situations in which testing is important, as mentioned above, but these are rarer.

There are no laboratories in Israel that perform plasma oxalate level testing. There are several laboratories, including the biochemistry laboratory at the Galilee Medical Center, that perform oxalate level testing in urine. Urine testing is performed as an initial screening in cases where hyperoxaluria is suspected and as part of the investigation of kidney stones.

Before PH1 medication was available, when the standard treatment was liver transplantation, it was customary to monitor only oxalate in urine in Israel. In the US and Europe, it was customary to monitor plasma oxalate levels after liver transplantation, and when the level dropped to close to normal, kidney transplantation was recommended. In situations where there was a liver and kidney donation from a deceased donor, it was not customary to delay the kidney transplant, and there were centers that performed dialysis for a certain period after liver-kidney transplantation while monitoring plasma oxalate levels. In Israel, as mentioned, it was not customary to perform dialysis after liver/liver-kidney transplantation, nor was it customary to monitor plasma oxalate levels after transplantation.

The situation changed after the new drug treatment was approved. Lumasiran was added to the Israeli health basket in 2022 for all PH1 patients. The treatment replaces liver transplantation, and as a result, there is a need to monitor plasma oxalate levels in the following situations3:

1. To monitor response to treatment with Lumasiran in dialysis patients who are not urinating (and therefore cannot be monitored for oxalate reduction in urine)
2. Prior to kidney transplantation in a PH1 patient with advanced renal failure treated with Lumasiran. According to current recommendations, plasma oxalate levels should be reduced to below 50 micromoles/liter prior to kidney transplantation.
3. After kidney transplantation in a patient treated with Lumasiran, to assess the risk and need for dialysis after transplantation in order to protect the kidney in case of high plasma oxalate levels.

Testing for oxalate in plasma is relatively more complicated than testing for oxalate in urine because urine levels are an order of magnitude higher than plasma levels (urine levels are measured in mmol/L and plasma levels in micromol/L), and the tests available on the market are more sensitive at higher concentrations. In addition, oxalate is unstable: ascorbic acid is converted to oxalate in a relatively basic environment (pH > 4), and therefore plasma must be acidified during test preparation.

The kit used to test for oxalate in urine in our biochemical laboratory is based on the enzyme oxalate oxidase and a color reaction (colorimetric) and is purchased from Biotech Trinity. According to the manufacturer's instructions, the kit is intended for testing oxalate levels in urine. This test is performed in our laboratory and has been internally validated according to the manufacturer's instructions.

There are two types of tests for plasma oxalate levels in laboratories around the world4 - mass spectrometry (gas or ion). The second method (mass spectrometry) is considered accurate for plasma oxalate but is quite expensive and not available to our laboratory. The use of the enzyme oxalate oxidase is accepted in research and for clinical purposes in leading laboratories around the world.

The biochemical laboratory at CHARITE Hospital in Berlin makes extensive use of plasma oxalate testing for clinical and research purposes. The laboratory and the nephrology department at CHARITE Hospital are considered world leaders in the field of hyperoxaluria. The director of the nephrology department at CHARITE, Prof. Felix Knopf, has published numerous articles on the subject, in which he used the enzymatic plasma oxalate test in the TRINITY kit6.

Given the need for plasma oxalate testing in Israel, and as we are a leading center in the field of hyperoxaluria in Israel, we are interested in making the test available in our institution's biochemical laboratory. In accordance with the means available to the laboratory here and after testing the effectiveness and reliability of the enzymatic test based on oxalate oxidase, we decided to validate the plasma oxalate test in our laboratory. Since the manufacturer intends the kit for urine testing only, it is not possible to perform validation based on the manufacturer's controls, and we needed external validation. In the pilot tests we have conducted so far, we have obtained acceptable values in accordance with the patient's clinical condition. Prof. Knopf from Charité Hospital in Berlin agreed to perform external validation for us for the plasma oxalate test performed in our biochemical laboratory.

Vitamin C (ascorbic acid) is a precursor to oxalate, so in situations where there is a tendency for high oxalate levels, such as hyperoxaluria and renal failure, it is recommended to avoid high doses of vitamin C supplements. KDOQI recommendations 2020 (Kidney Disease Outcome Quality Initiative)7 regarding vitamin C supplements in patients with stage 1-5 chronic kidney disease is to give a relatively low dose to patients at increased risk of vitamin C deficiency while monitoring oxalate levels or the development of calcium oxalate stones in the kidney. Previous studies have shown a link between vitamin C supplements or ascorbic acid levels and oxalate levels in patients with chronic renal failure and dialysis patients8,9. Low vitamin C levels are associated with the relatively poor nutritional status of patients with renal failure and may manifest clinically with symptoms of vitamin C deficiency. The dialysis unit at the Galilee Medical Center described a case of a dialysis patient who suffered from symptomatic vitamin C deficiency that required treatment with high doses of oral vitamin C. High blood oxalate levels in dialysis patients have been found to be associated with a higher incidence of cardiovascular complications. Hence the recommendations to exercise caution when administering vitamin C supplements in cases of renal failure or dialysis, where oxalate clearance by the kidneys is poor and therefore oxalate produced from excess ascorbic acid may accumulate in the blood and various tissues in the body and cause multi-system damage.

There are few studies that have examined the relationship between oxalate levels and vitamin C levels in various degrees of renal failure and hyperoxaluria. We are interested in testing vitamin C levels in addition to plasma oxalate levels for all participants in the above study in order to assess vitamin C deficiency in the population of patients with renal failure or hyperoxaluria and to assess the relationship between vitamin C levels and blood oxalate levels in this group.

Main objective - validation of plasma oxalate level testing Additional objective - examination of the relationship between vitamin C levels and plasma oxalate levels in patients with renal failure and hyperoxaluria treated with Lumicran.

Importance of conducting the research:

1. Establishment of a laboratory service that does not currently exist in Israel and is clinically important for treatment decisions, as detailed above.
2. Assessing the relationship between vitamin C levels and oxalate levels in a population of patients with renal failure and hyperoxaluria will help in the tailored treatment of these patients and in preventing complications of vitamin C deficiency on the one hand, or hyperoxaluria secondary to vitamin C excess on the other.

Methods:

Number of samples:

1. For the validation test, 30 blood samples will be taken from 30 different patients. The samples will be taken from a variety of patients in order to obtain a wide range of plasma oxalate levels. Approximately 5 samples will be taken from healthy volunteers, approximately 20 samples from dialysis patients with no history of hyperoxaluria, and approximately 5 samples from hyperoxaluria patients receiving medication or who have undergone liver transplants.

   Each sample will be sent for oxalate level testing at the biochemical laboratory at the Galilee Medical Center + biochemical laboratory at the Charité Hospital in Berlin + vitamin C level testing at Sheba Hospital.
2. To examine the relationship between vitamin C levels and oxalate levels in dialysis patients: approximately 20 additional blood samples will be taken from dialysis patients, and oxalate levels will be tested at the local laboratory and vitamin C levels at the Sheba Medical Center laboratory, Tel Aviv, Israel.

Total number of participants: 50 Oxalate plasma testing protocol - attached in the appendix. The protocol has been approved by the laboratory where the external validation will be performed.

Each sample will undergo immediate centrifugation, and the plasma will be divided into two test tubes and stored frozen (-80°C). One test tube will be sent for testing at the laboratory in Berlin, and one test tube will remain here and be tested at our laboratory.

The sample handling stage until freezing is the same as it will be performed here.

The sample handling process in the laboratory here will be performed by one laboratory employee.

The samples will be sent frozen to the laboratory in Berlin. Stage two - sample processing after thawing - will be carried out according to a protocol agreed upon by both laboratories in order to prevent differences in sample processing. We will also coordinate the days on which the tests are carried out between the two laboratories in order to prevent differences resulting from the duration of sample preservation in frozen storage.

The protocol was jointly written by us and the laboratory in Berlin. Vitamin C level testing will be performed at an external laboratory (Sheba).

Statistics - After receiving the test results from Berlin, we will compare the results obtained there and here using the following tests:

Quantitative data will be described using means and standard deviations, median, interquartile range (IQR), and range.

Paired sample comparison tests - To examine the differences between two paired samples using a paired sample T test (if the differences are normally distributed) or a Wilcoxon signed rank test if the distribution of the differences is not normal. A 95% confidence interval will be calculated for the difference between the paired samples.

Correlation tests - to examine the relationship between the paired samples. Pearson's correlation coefficient test or alternatively Spearman's correlation coefficient test (selected according to sample size and distribution shape) Bland-Altman plots and scatter plots will be used to illustrate the differences between the results.

A P value lower than 5% will be considered statistically significant. Anonymity: Samples will be marked with a code provided here, without identifying details on the forms or test tubes. The coding table will be kept separately on the principal investigator's computer and in a separate binder in the research coordinator's cabinet.

Informed consent: Volunteers will sign an informed consent form after receiving an explanation of the significance of the test.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent

Exclusion Criteria:

* Not willing to participate

Ages: 1 Minute to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy patients Dialysis patients without a background of hyperoxaluria Hyperoxaluria patients receiving drug treatment or after a liver transplant Patients with advanced kidney failure not on dialysis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
correlation of plasma oxalate between local and external laboratories | 1 year
  The plasma oxalate results from local and external laboratories will be compared by statistical analysis:
  Comparison tests for paired samples - to examine the differences between two paired samples using the paired sample T test or the Wilcoxon signed rank test if the distribution of the differences is not normal. A 95% confidence interval will be calculated for the difference between the paired samples.
  Correlation tests -Pearson's correlation coefficient test or alternatively Spearman's correlation coefficient test Bland-Altman plot and Scatter plot curves will be used to demonstrate the difference between the results.
  A P value lower than 5% will be considered statistically significant. The investigators aim to to have non significant differences between the results of the laboratories in order to conclude that the results in the local laboratory are valid.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfau A, Ermer T, Coca SG, Tio MC, Genser B, Reichel M, Finkelstein FO, Marz W, Wanner C, Waikar SS, Eckardt KU, Aronson PS, Drechsler C, Knauf F. High Oxalate Concentrations Correlate with Increased Risk for Sudden Cardiac Death in Dialysis Patients. J Am Soc Nephrol. 2021 Sep;32(9):2375-2385. doi: 10.1681/ASN.2020121793. Epub 2021 Jul 19. PMID 34281958
- [Background] Ikizler TA, Burrowes JD, Byham-Gray LD, Campbell KL, Carrero JJ, Chan W, Fouque D, Friedman AN, Ghaddar S, Goldstein-Fuchs DJ, Kaysen GA, Kopple JD, Teta D, Yee-Moon Wang A, Cuppari L. KDOQI Clinical Practice Guideline for Nutrition in CKD: 2020 Update. Am J Kidney Dis. 2020 Sep;76(3 Suppl 1):S1-S107. doi: 10.1053/j.ajkd.2020.05.006. PMID 32829751
- [Background] Stokes F, Acquaviva-Bourdain C, Hoppe B, Lieske JC, Lindner E, Toulson G, Vaz FM, Rumsby G. Plasma oxalate: comparison of methodologies. Urolithiasis. 2020 Dec;48(6):473-480. doi: 10.1007/s00240-020-01197-4. Epub 2020 May 29. PMID 32472220
- [Background] Ladwig PM, Liedtke RR, Larson TS, Lieske JC. Sensitive spectrophotometric assay for plasma oxalate. Clin Chem. 2005 Dec;51(12):2377-80. doi: 10.1373/clinchem.2005.054353. No abstract available. PMID 16306102
- [Background] Oka Y, Miyazaki M, Matsuda H. Plasma Oxalate Concentration and Patients With CKD. Kidney Int Rep. 2021 Mar 1;6(4):1194. doi: 10.1016/j.ekir.2020.10.041. eCollection 2021 Apr. No abstract available. PMID 33912770